CLINICAL TRIAL: NCT00158496
Title: Clinical Trial of the Efficacy of the Combination of Pegylated Interferon (PEG-IFNα-2a) Plus Ribavirin in Egyptian Patients With Untreated Chronic Hepatitis C
Brief Title: Chronic Hepatitis C Treatment by Pegylated Interferon and Ribavirin in Naive Egyptian Patients (ANRS 1211)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 1211
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2007-04-24 (Estimated); Status verified 2007-04

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic Hepatitis C; Genotype 4; Pegylated Interferon; Ribavirin; Egypt
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: pegylated interferon alpha2a
Drug: ribavirin

SUMMARY:
Chronic hepatitis C is a liver disease related to a virus: hepatitis C virus (HCV). The type of HCV present in Egypt (genotype 4), has the reputation to respond poorly to Interferon treatment at the chronic stage. Pegylated Interferon is a new form of Interferon that stays in the body for longer time and allows the patient to take less injection per week. It has proved to be more effective than standard Interferon. The combination of two drugs, Interferon and Ribavirin, is considered to be the best treatment available for chronic hepatitis C.

DETAILED DESCRIPTION:
Egypt is the country with the highest HCV prevalence worldwide, and the number of infected Egyptians is estimated around 8 million. The HCV genotype circulating in Egypt is genotype 4. This genotype has the reputation, based on the few available data, to respond poorly to treatment. This study will estimate the safety and efficacy of the combination of peg-IFNα-2a plus Ribavirin, in Egyptian patients with chronic hepatitis C. This treatment has been chosen based on its better expected efficacy compared to pegylated interferon alone.

The primary objective of the study is to assess the efficacy and tolerance of the combination of pegylated interferon (peg-IFNα-2a) plus ribavirin in Egyptian patients with chronic hepatitis C and with no prior treatment for HCV.

Methods: Open trial. Follow-up duration: 72 weeks. Enrolment duration: 18 months. Total trial duration: 3 years and a half, including trial analysis (carried out in the 6 months following the follow-up completion of the last patient). Total number of patients: 100. Precision around the expected efficacy rate (40% in intention-to-treat analysis): 9.6%.

Treatment strategy: Peg-IFNα-2a 180microg/week for 48 weeks, Ribavirin at least 11 mg/kg/day for 48 weeks Main inclusion criteria: HCV RNA positive by PCR; METAVIR score : >A2 and >= F1 or >= A1 and > F2; ALAT over 1.5*N; no prior treatment with IFNalpha, PEG-IFNalpha and ribavirin Main exclusion criteria : Liver disease other than hepatitis C; advanced liver disease; negative HCV RNA.

Patient from a cohort follow-up conducted in a village in rural Egypt with High HCV prevalence (Menoufia governorate) will be proposed to participate in the trial. Pre-enrolment investigations, liver biopsy, and patients follow-up will be carried out at a local hospital. Blood test analyses will be carried out under the responsibility of Hepatitis Virology Reference Laboratory at the National Hepatology and Tropical Medicine Institute, Cairo; trial monitoring will be carried out by the Department of Community Medicine of Ain Shams; methodological assistance from the "Unite des Maladies Emergentes" at Pasteur Institute and INSERM U444, Paris.

Treatment for patients with HCV RNA by qualitative PCR still positive after 24 weeks of the combination Peg-IFNα-2a with ribavirin, will be stopped.

ELIGIBILITY:
Inclusion Criteria:

* HCV antibodies using a third generation test
* HCV RNA positive by PCR
* Liver biopsy in the past 18 months with METAVIR score over A2 and over or equal to F1, or over or equal A1 and over F2
* ALT over 1.5 time the normal range in the 24 weeks prior to inclusion (Week-28; W-2);
* Patients never treated with ribavirin, IFNalpha or PEG-IFNalpha
* Normal albumin
* Prothrombin time over or equal to 60 percent
* Normal bilirubin
* Alpha-foeto-protein under or equal to 3 times the normal range for the laboratory
* HBs antigen negative
* Two negative Kato test (for S.mansoni) three days apart
* Hemoglobin over or equal 11g/dl,
* Leucocytes over or equal 3000/mm3
* Neutrophils over or equal 1500/mm3
* Platelets over or equal 100 000/mm3
* Blood creatinin over or equal 150 micromol/l
* Normal TSH
* Anti-nuclear antibodies under 1/160
* Fasting blood sugar between 70-115mg/dl (if glucose intolerance or diabetes: HbA1C <= 8,5%)
* Normal ophthalmologic examination in patients with history of blood pressure and/or diabetes
* Effective contraception during the treatment period
* No breastfeeding during the study period.
* Signed informed consent

Exclusion Criteria:

* Co-infection with hepatitis B (positive HBs antigen)
* Hemochromatosis
* Alpha-1 anti-trypsin deficiency
* Wilson disease
* Alcoholism-related liver disease
* Gilbert disease
* Alcohol intake over 50g/day for males and 40 g/day for females
* Ongoing intravenous drug use
* Aggravated liver cirrhosis (history or presence of ascitis, oesophageal varicosis, liver encephalopathy)
* Hepatocellular carcinoma
* Psychiatric disease: history of severe nervous breakdown or severe psychiatric diseases such as major psychosis, suicidal ideas, suicide attempts…
* Epilepsy
* Auto-immune disease
* Heart disease in the six months preceding enrolment - patients with significant changes at EKG
* Uncontrolled diabetes
* Chronic respiratory insufficiency with hypoxemia <10 kPa
* Medical or surgical condition, non-stabilised, with life expectancy lower than two years.
* Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2002-08; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
- Disappearance of HCV RNA by qualitative PCR 24 weeks after the end of treatment

SECONDARY OUTCOMES:
Evaluation of HCV RNA at 12 and 24 weeks
changes in HCV RNA load during treatment
Normalization of ALT during treatment and 24 weeks after the end of treatment
Study of side effects
Histological changes 24 weeks after the end of treatment (decrease by at least 1 point of the Metavir score)

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Fontanet, Study Chair — Institut Pasteur de Paris; Mostafa K Mohamed, Principal Investigator — National Hepatology and Tropical Medicine Research Institute
Locations (2):
- Egypt (2):
  - Ismail Sallam hospital, Zawiat Razin, Menoufia
  - National Hepatology and Tropical Medicine Research Institute, Cairo

REFERENCES:
- [Background] Marzouk D, Sass J, Bakr I, El Hosseiny M, Abdel-Hamid M, Rekacewicz C, Chaturvedi N, Mohamed MK, Fontanet A. Metabolic and cardiovascular risk profiles and hepatitis C virus infection in rural Egypt. Gut. 2007 Aug;56(8):1105-10. doi: 10.1136/gut.2006.091983. Epub 2006 Sep 6. PMID 16956918
- [Background] Mohamed MK, Bakr I, El-Hoseiny M, Arafa N, Hassan A, Ismail S, Anwar M, Attala M, Rekacewicz C, Zalata K, Abdel-Hamid M, Esmat G, Fontanet A. HCV-related morbidity in a rural community of Egypt. J Med Virol. 2006 Sep;78(9):1185-9. doi: 10.1002/jmv.20679. PMID 16847958
- [Background] Bakr I, Rekacewicz C, El Hosseiny M, Ismail S, El Daly M, El-Kafrawy S, Esmat G, Hamid MA, Mohamed MK, Fontanet A. Higher clearance of hepatitis C virus infection in females compared with males. Gut. 2006 Aug;55(8):1183-7. doi: 10.1136/gut.2005.078147. Epub 2006 Jan 24. PMID 16434426
- [Background] Arafa N, El Hoseiny M, Rekacewicz C, Bakr I, El-Kafrawy S, El Daly M, Aoun S, Marzouk D, Mohamed MK, Fontanet A. Changing pattern of hepatitis C virus spread in rural areas of Egypt. J Hepatol. 2005 Sep;43(3):418-24. doi: 10.1016/j.jhep.2005.03.021. PMID 16019104
- See also: Sponsor web page - information in french and english — http://www.anrs.fr